CLINICAL TRIAL: NCT00081614
Title: A Phase II, Multicenter, Randomized, Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of Tarceva (Erlotinib Hydrochloride) in Combination With Avastin (Bevacizumab) Versus Avastin Alone for Treatment of Metastatic Renal Cell Carcinoma
Brief Title: A Study Evaluating Tarceva in Combination With Avastin Versus Avastin Alone in Treating Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVF2938g; NCT00091221 (obsolete NCT alias)
Record Dates: First submitted 2004-04-15; First posted 2004-04-20 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Renal Cell Carcinoma; Metastases
Keywords: Metastatic renal cell carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Bevacizumab; Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Avastin (bevacizumab)
Drug: Tarceva (erlotinib HCl)

SUMMARY:
The primary purpose of the study is to assess the potential benefit of combining two targeted therapies (an anti-EGF inhibitor along with an anti-VEGF inhibitor). The goal will be to determine whether the addition of Erlotinib to Avastin will improve the benefit in metastatic renal cell carcinoma (RCC) with regard to time to progression, response rate, duration of response, and survival compared with Avastin alone. Since Avastin has been shown to be active in renal cancer, the goal will be to assess whether this activity can be enhanced with Erlotinib.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically confirmed RCC of clear cell histology
* Confirmed metastatic RCC
* Age >=18 years
* ECOG performance status of 0 or 1
* Life expectancy >=3 months
* Prior nephrectomy
* Measurable disease, as defined by RECIST
* Use of an acceptable means of contraception (potentially fertile men and women)

Exclusion Criteria:

* RCC with predominantly sarcomatoid features
* Prior systemic or adjuvant therapy for RCC
* Prior radiotherapy for RCC within 28 days prior to Day 0, with the exception of single fraction radiotherapy given for the indication of pain control
* Treatment with Avastin, Tarceva, or other agents, either investigational or marketed, that act by either EGFR inhibition or anti-angiogenesis mechanisms
* 24-hour urine collection with >=1 g of protein
* INR >=1.5, except for subjects receiving warfarin therapy
* Serum creatinine >2.0 mg/dL
* Serum calcium >10 mg/dL (corrected)
* Absolute neutrophil count (ANC) <1500/uL
* Platelet count <75,000/uL
* Total bilirubin >2.0 mg/dL
* AST or ALT >5× the upper limit of normal (ULN) for subjects with documented liver metastases; >2.5 × ULN for subjects without evidence of liver metastases
* LDH >1.5× ULN
* Hemoglobin <9 gm/dL (may be transfused or receive epoetin alfa [e.g., Epogen] to maintain or exceed this level)
* History of serious systemic disease, including myocardial infarction within the last 6 months, uncontrolled hypertension (blood pressure >160/110 mmHg on medication), unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia, are eligible), or Grade II or greater peripheral vascular disease
* History of acute stroke within 6 months prior to randomization
* Patients on dialysis
* Other invasive malignancies, including bladder cancer and low-grade endometrial cancer, within 5 years of randomization (other than squamous or basal cell carcinoma of the skin)
* Pregnancy or breast feeding
* Inability to comply with study and/or follow-up procedures
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* History or clinical evidence of central nervous system or brain metastases
* History of bowel or gastric perforation
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure during the course of the study

  * Fine needle aspirations or core biopsies within 7 days prior to Day 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Bay Area Cancer Research Group, Concord, California
  - UCLA School of Medicine, Los Angeles, California
  - Kaiser Permanente Medical Group, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - UCHSC - Urologic Oncology, Aurora, Colorado
  - Bennett Cancer Center, Stamford, Connecticut
  - Lynn Regional Cancer Center - West, Boca Raton, Florida
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Wayne State University / Harper University Hospital, Detroit, Michigan
  - St. Joseph Oncology, Saint Joseph, Missouri
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - NYU School of Medicine, New York, New York
  - Our Lady of Mercy Medical Center, The Bronx, New York
  - Northwestern Carolina Oncology & Hematology, Hickory, North Carolina
  - Raleigh Hematology Oncology, Raleigh, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Bukowski RM, Kabbinavar FF, Figlin RA, Flaherty K, Srinivas S, Vaishampayan U, Drabkin HA, Dutcher J, Ryba S, Xia Q, Scappaticci FA, McDermott D. Randomized phase II study of erlotinib combined with bevacizumab compared with bevacizumab alone in metastatic renal cell cancer. J Clin Oncol. 2007 Oct 10;25(29):4536-41. doi: 10.1200/JCO.2007.11.5154. Epub 2007 Sep 17. PMID 17876014
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227